CLINICAL TRIAL: NCT00960882
Title: Gastric Tolerability and Pharmacokinetics of DMMET-01. Daily Intake for 30 Days, in Normal Alimentation Conditions, in Healthy Volunteers.
Brief Title: Gastric Tolerability and Pharmacokinetics of DMMET-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMMET 1011/07
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Diabetes; gastric tolerability
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DMMET-01 (Experimental)
  Interventions: Drug: DMMET-01

INTERVENTIONS:
Drug: DMMET-01 — 1050.6 mg daily for 30 days

SUMMARY:
The purpose of this study is to determine the gastric tolerability and the pharmacokinetics of a new drug for the treatment of type 2 diabetes, DMMET-01, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Mexican healthy subjects with normal clinical laboratory test results and imaging (hematology, blood chemistry, urine test, VDRL, Hepatitis B, HIV, chest radiography and electrocardiogram)

Exclusion Criteria:

* Familiar or personal history of diabetes
* History of drug or alcohol abuse within the 2 years prior to the study
* A smoking habit greater tha 10 cigarettes per day
* Intercurrent disease
* Intercurrent treatment with any drug

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
DMMET-01 Plasmatic concentration | 48 hrs (7.5; 15; 30; 45; 60; 75; 90; 120; 150; 180; 205; 240; 360; 480; 600; 720; 1440 and 2880 min)

SECONDARY OUTCOMES:
Lanza score | 30 days (0 and 30)
plasmatic glucose | 24 hours (6,12,18 and 24)
glycated hemoglobin | 24 hours (0 and 24)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Torres, PhD, Principal Investigator — UANL, Pharmacology and toxicology department; Jorge A Gonzalez, Master, Study Director — Laboratorios Silanes S.A. de C.V.
Locations (1):
- Pharmacology and toxicology department, UANL, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided